CLINICAL TRIAL: NCT07196917
Title: Prospective Cohort of Integrated Traditional Chinese and Western Medicine in China
Status: Not yet recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Hubei College of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Hubei Provincial Center for Disease Control and Prevention (Other); Wuhan Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Long Pin Pin, lecturer, Huazhong University of Science and Technology
Other Study IDs: 2023ZD0S09900)
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Respiratory Tract Diseases; Cancer; Endocrine System Diseases; Death
MeSH Terms: conditions — Cardiovascular Diseases; Respiratory Tract Diseases; Neoplasms; Endocrine System Diseases; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To further explore the application prospects of integrated Traditional Chinese and Western medicine in chronic disease prevention and control and health management, this study intends to establish a large, prospective, integrated Traditional Chinese and Western medicine cohort in Hubei Province. This study will conduct long-term follow-up and multi-dimensional data collection to systematically reveal the associations between Traditional Chinese Medicine (TCM) constitution types and chronic diseases, the aging process, and multi-morbidity, thereby developing an integrated health management strategy with local characteristics. This study will fill the current gap in systematic evidence linking TCM constitutions to the prevalence of modern diseases, providing a solid demographic and biological foundation for the integrated development of Traditional Chinese and Western medicine. It will also contribute to meeting the needs for early disease warning, early intervention, and personalized care under the "Healthy China" strategic goal.

ELIGIBILITY:
Inclusion Criteria:

Age: Participants aged 30 to 74 years

Physical Functionality: Free from severe physical disabilities impacting mobility or communication, with preserved ability to comprehend and respond to study procedures

Informed Consent: Capable of providing written informed consent voluntarily after receiving full study disclosure

Exclusion Criteria:

Residents living in functional areas (e.g., work sheds, military units, student dormitories, nursing homes, etc.)

Individuals unable to communicate normally

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Targeting urban and rural residents across multiple regions in Hubei Province, this study plans to recruit 1 million participants. Standardized protocols will be employed for baseline questionnaire surveys, physical examinations, and biological sample collection.
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prospective Cohort of Integrated Traditional Chinese and Western Medicine in China | From enrollment to the 10-year follow-up
Incidence of major chronic diseases (coronary heart disease, stroke, diabetes, COPD, lung cancer, colorectal cancer, gastric cancer, liver cancer, and esophageal cancer) | From baseline (enrollment) to 10-year follow-up Measurement Tool: Standardized physician-adjudicated diagnosis based on ICD-10 codes, confirmed through hospital electronic medical records and disease registries

SECONDARY OUTCOMES:
All-cause mortality | From baseline to 10-year follow-up
  Time Frame: From baseline to 10-year follow-up Measurement Tool: Death registry linkage and hospital records Unit of Measure: Mortality rate per 1,000 person-years

OTHER OUTCOMES:
Cause-specific mortality (cardiovascular, cancer, respiratory, metabolic) | From baseline to 10-year follow-up
  Time Frame: From baseline to 10-year follow-up Measurement Tool: Death registry and ICD-10 coded cause of death Unit of Measure: Mortality rate per 1,000 person-years
Prevalence and progression of multimorbidity (≥2 chronic conditions) | Baseline to 10-year follow-up
  Time Frame: Baseline to 10-year follow-up Measurement Tool: Questionnaire survey and physician-adjudicated diagnosis using ICD-10 Unit of Measure: % of participants with multimorbidity